CLINICAL TRIAL: NCT07078643
Title: Comparison of the Effects of Superior Hypogastric Plexus Block and Erector Spinae Plane Block on Postoperative Analgesia in Total Laparoscopic Hysterectomy Surgery
Brief Title: Comparison of the Effects of Blocks on Postoperative Analgesia in Total Laparoscopic Hysterectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MACİD ORDU, Assistant Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DrLutfiKirdarTRH-MO-01
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Total Laparoscopic Hysterectomy
Keywords: Postoperative Pain; Erector Spinae Plane Block; Superior Hypogastric Plexus Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: "This study uses a parallel design where participants are randomly assigned to one of three groups: Superior Hypogastric Plexus Block (SHPB), Erector Spinae Plane Block (ESPB), or Control group. Each group receives its respective intervention or no block in the control group. Outcomes are measured postoperatively to compare analgesic efficacy among groups."
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study was conducted in a double-blind manner. Participants, care providers performing the block procedures, and outcome assessors were blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Superior Hypogastric Plexus Block (SHPB) Group (Active Comparator): SHPB Group: In this group, patients received a superior hypogastric plexus block (SHPB) following total laparoscopic hysterectomy. After uterus removal and vaginal cuff closure, and before trocar removal, the injection site was identified laparoscopically. The block was performed in all patients by a single surgeon experienced in SHPB.
  Interventions: Procedure: Superior Hypogastric Plexus Block (SHPB)
- Erector Spinae Plane Block Group (Active Comparator): ESPB Group: Patients in this group received erector spinae plane block (ESPB) during anesthesia maintenance after surgery. Patients were positioned in the lateral decubitus position. At the T10 level, the ultrasound probe was placed in the midline to identify spinous processes, then moved 2-3 cm laterally to visualize the transverse process, trapezius, and erector spinae muscles. The same procedure was performed on the opposite side. All blocks were performed by a single anesthesiologist experienced in ESPB.
  Interventions: Procedure: Erector Spinae Plane Block (ESPB)
- Control Group (No Intervention): Control Group: Patients in this group did not receive any block and were managed with standard postoperative care only. This group served as the comparison group to evaluate the effects of the block interventions.

INTERVENTIONS:
Procedure: Superior Hypogastric Plexus Block (SHPB) — Laparoscopic superior hypogastric plexus block with bupivacaine and lidocaine injection near sacral promontory.
  Arms: Superior Hypogastric Plexus Block (SHPB) Group
Procedure: Erector Spinae Plane Block (ESPB) — Erector spinae plane block with ultrasound-guided injection of bupivacaine and lidocaine at T10 level.
  Arms: Erector Spinae Plane Block Group

SUMMARY:
Total laparoscopic hysterectomy (TLH) is one of the most commonly performed gynecological surgeries today. Various analgesic techniques are used for the management of postoperative pain. The aim of this study is to compare the postoperative analgesic efficacy of superior hypogastric plexus block (SHPB) and erector spinae plane block (ESPB) in patients undergoing TLH procedures.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, single-center clinical trial aims to compare the postoperative analgesic efficacy of Superior Hypogastric Plexus Block (SHPB) and Erector Spinae Plane Block (ESPB) in patients undergoing total laparoscopic hysterectomy (TLH).

Following ethics committee approval (2022/514/220/10), the study was conducted between March 2022 and March 2023. Patients aged 18 to 65 years, classified as ASA physical status I-II and scheduled for elective TLH, were enrolled. Participants were randomly assigned into three groups using computer-generated randomization (n=30 per group): SHPB, ESPB, and Control. Both the anesthesiologist performing postoperative evaluations and the patients were blinded to group allocation.

All patients received general anesthesia in accordance with a standardized protocol.

ESPB was performed bilaterally at the T10 level under ultrasound guidance. SHPB was performed laparoscopically at the L5-S1 level after uterine removal. No regional block was applied in the control group.

Postoperative pain management was provided to all patients via patient-controlled analgesia (PCA). Pain levels were evaluated using the Visual Analog Scale (VAS) at postoperative 0, 30, 60, 90, and 120 minutes, and at 6, 12, and 24 hours.

This study aims to investigate whether SHPB provides more effective visceral analgesia compared to ESPB and whether this leads to reduced opioid requirements and improved patient satisfaction following TLH.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 65 years
* Scheduled for elective total laparoscopic hysterectomy (TLH)
* Classified as American Society of Anesthesiologists (ASA) physical status I or II
* Able to provide written informed consent in accordance with the Declaration of Helsinki

Exclusion Criteria:

* Refusal to participate or inability to provide informed consent
* Body mass index (BMI) ≥ 35 kg/m²
* Inability to cooperate or follow instructions
* Presence of spinal or paravertebral deformity
* Known coagulopathy or use of anticoagulant therapy
* Known hypersensitivity or allergy to local anesthetic drugs used in the study
* Requirement for postoperative intensive care
* History of chronic opioid use (longer than four weeks prior to surgery)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Total Tramadol Consumption | Postoperative 0-24 hours
  The total amount of tramadol administered via a patient-controlled analgesia (PCA) device within the first 24 hours after total laparoscopic hysterectomy. This measurement is used to compare the postoperative analgesic efficacy of superior hypogastric plexus block (SHPB) and erector spinae plane block (ESPB) with the control group receiving no block. Tramadol consumption is recorded in milligrams (mg) and extracted directly from PCA device logs.

SECONDARY OUTCOMES:
Postoperative Pain Intensity (VAS Scores) | Postoperative 0-24 hours
  Pain levels will be measured using the Visual Analog Scale (VAS), a 10 cm horizontal line labeled "no pain" at 0 cm and "worst imaginable pain" at 10 cm. Patients will indicate their pain intensity at postoperative time points (e.g., 1h, 6h, 12h, 24h). The score is determined by measuring the distance in centimeters from the "no pain" anchor to the patient's mark. Higher scores indicate greater pain intensity.
Time to First Rescue Analgesia | Postoperative 0-24 hours
  Duration from the end of surgery to the time the patient first requests additional analgesia beyond the standard postoperative regimen.
Incidence of Postoperative Nausea and Vomiting (PONV) | Postoperative 0-24 hours
  The proportion of patients experiencing nausea and/or vomiting within the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Macid Ordu, MD, Principal Investigator — Kartal Dr. Lütfi Kırdar Training and Research Hospital
Locations (1):
- Kartal Dr. Lütfi Kırdar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data due to institutional data protection policies and ethical considerations related to participant privacy.